CLINICAL TRIAL: NCT05440357
Title: Second-line Pharmacotherapy Patterns and Outcomes of Advanced Gastrointestinal Stromal Tumor: A Real-world Study
Status: Recruiting | Type: Observational
Sponsor: Xinhua Zhang, MD (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Peking University Shenzhen Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); Hainan Cancer Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); Yunnan Cancer Hospital (Other); Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Xinhua Zhang, MD, First Affiliated Hospital, Sun Yat-Sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: No.[2021]784
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, multicenter, observational real-world study to explore the second-line Pharmacotherapy patterns and clinical outcomes in GIST patients who progressed on or were intolerant to first-line anticancer treatment.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Gastrointestinal stromal tumors (GIST) are thought to develop from the interstitial cells of Cajal or their stem cell precursors. They are the most common mesenchymal tumors occurring in the gastrointestinal (GI) tract. The annual incidence of GIST is about 1/100,000 ~ 2/100,000 globally. Previous data showed that the incidence of GIST was 0.43 per 100,000 in Shanxi Province and 2.11per 100,000 in Shanghai in China.

Surgery is the primary therapy for patients with localized resectable disease. GIST that is metastatic or locally advanced but unresectable is treated with tyrosine kinase inhibitors (TKIs) that target KIT or PDGFRA.

Imatinib is recommended as the first-line standard treatment for metastatic or unresectable advanced GIST. Most patients with initial clinical benefits from Imatinib eventually progress. However, approximately 10% -14% of GIST is primarily resistant to imatinib and 90% of patients will develop secondary drug resistance within 4 years with imatinib treatment.

For patients who failed imatinib first-line treatment, Sunitinib is the standard second-line therapy but not the optimal treatment regimen in clinical practice. Other TKIs targeting KIT is also used in the second-line setting. A phase 3 study to evaluate sunitinib's efficacy in advanced GIST compared with placebo, showed that the mPFS was 5.6 months [2], while a phase I study of ripretinib demonstrated that the mPFS was10.7months as a second-line treatment in advanced GIST[4]. Another single-arm second-line treatment study of dasatinib also suggested that dasatinib had a tumor suppression effect in the treatment of advanced GIST with imatinib treatment failure, with mPFS of 2.9 months, and mOS of 19 months, especially for patients with SRC overexpression and PDGFRA D842V mutation [5]. There is a lack of real-world data on advanced GIST patients who have progressed on first-line treatment with different treatment patterns, and the benefits are also unknown.

The investigators initiate this prospective, observational, real-world study that aims to explore the second-line treatment patterns and the clinical outcomes in GIST patients who progressed on or were intolerant to first-line treatment in real-world clinical practice.

STUDY PROCEDURE Approximately 100 patients will be enrolled. According to the inclusion criteria, patients will receive second-line treatment that was recommended by the current guidelines, including sunitinib, imatinib dose-escalation, repritinib, dasatinib, and other drugs based on the physician's judgment. Data will be collected based on a real-world setting.

SCREENING PERIOD During the screening period, the informed consent form will be signed before enrolling. Radiologic imaging and dermatologic examination should be performed within 30 days before the first day of enrollment. Baseline information, including medical history, previous treatment pattern, ECOG PS score, EORTC-QLQ-C30 scale, molecular detection, and any laboratory test should be recorded.

OBSERVATION PERIOD Patients will be enrolled in the study after confirmation of all eligibility criteria. The treatment patterns will be decided by the physician. Study visits during the Treatment Period will occur every 2 months. Regular physical examination, vital signs, imaging examination, tumor assessment(PFS and ORR), EORTC-QLQ-C30, 2. ECOG PS score, the dose of drug and dose Administration, and drug-related adverse events will be recorded during each visit.

FELLOW-UP PERIOD Patients will be contacted by phone call for the Safety Follow-up Visit 30 days after the last visit of study. Any AEs, medications, including anticancer treatments, and survival status will be followed during this period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged ≥ 18 years.
* Patients who have histologically confirmed metastatic or unresectable GIST.
* Patients who received imatinib at a fixed dose or 1 other TKI as prior treatment regimens. Patients who experienced intolerance to prior therapies must have objective disease progression before enrollment.
* Patients must have at least a measurable lesion according to mRECIST Version 1.1.
* According to the current GIST national guidelines, patients who receive second-line treatments, including but not limited to sunitinib, imatinib dose escalation, ripretinib, dasatinib, and other drug treatments.
* Patients with an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2 at screening.

Exclusion Criteria:

* Patients who previously received two or more TKIs as prior treatment regimens.
* Patients with a life expectancy of fewer than three months.
* Patients who are pregnant and lactating.
* Patients with an estimated poor adherence or inability to complete follow-up.
* Patients who are not appropriate to enroll due to the investigator's consideration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 100 patients with metastatic or unresectable advanced gastrointestinal stromal tumors from tier-3 hospitals who meet the criteria will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 1 year
  The primary objective is to demonstrate the proportion of patients with progression-free survival (PFS) determined by radiological assessment per modified Response Evaluation Criteria in Solid Tumors (mRECIST), version 1.1 in patients with advanced GIST following the second-line treatment.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  To evaluate PFS determined by radiology assessment per mRECIST, version 1.1 in patients with advanced GIST treated with second-line treatment.
overall survival (OS) | 2 years
  To evaluate overall survival (OS) in patients with advanced GIST treated with second-line treatment.
objective response rate (ORR) | 2 years
  To evaluate objective response rate (ORR) determined by radiology assessment per mRECIST, version 1.1 in patients with advanced GIST treated with second-line treatment.
Time to objective response | 1 year
  Time to objective response is defined as the interval between the date of randomization and the earliest documented evidence of the best objective reponse based on the independent radiologic review the best objective response rate (ORR) determined by radiology assessment per mRECIST, version 1.1 in patients with advanced GIST treated with second-line treatment.
R0/R1 resection rate | 2 years
  To evaluate the proportion of patients who performed R0/R1 resection surgery with advanced GIST treated with second-line treatment.
EORTC QLQ-C30 | Difference between baseline and every 3 month during the follow-up period
  QOL as measured by using EORTC QLQ-C30, Change in Individual Scores in Patients With Advanced GIST Treated under second-line treatment
Safety-TEAEs | 2 years
  Treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), serious adverse events (SAEs), dose reduction or discontinuation of study drug due to toxicity; changes from baseline in ECOG PS; Incidence of surgical complications.

OTHER OUTCOMES:
To explore the association of cilinical outcomes with treatment pattern | 2 years
  To evaluate the association of cilinical outcomes with baseline genotype mutation status,treatment parrern, R0/R1 resection status

CONTACTS AND LOCATIONS:
Overall Officials: zhang xinhua, PhD, Principal Investigator — First affiliated hosptial,Sun Yat-sen university
Locations (8):
- China (8):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The first affiliated hospital,Sun yat-sen university, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Hainan Cancer Hospital, Haikou, Hannan
  - Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi

REFERENCES:
- [Background] Demetri GD, van Oosterom AT, Garrett CR, Blackstein ME, Shah MH, Verweij J, McArthur G, Judson IR, Heinrich MC, Morgan JA, Desai J, Fletcher CD, George S, Bello CL, Huang X, Baum CM, Casali PG. Efficacy and safety of sunitinib in patients with advanced gastrointestinal stromal tumour after failure of imatinib: a randomised controlled trial. Lancet. 2006 Oct 14;368(9544):1329-38. doi: 10.1016/S0140-6736(06)69446-4. PMID 17046465
- [Background] Li J, Gao J, Hong J, Shen L. Efficacy and safety of sunitinib in Chinese patients with imatinib-resistant or -intolerant gastrointestinal stromal tumors. Future Oncol. 2012 May;8(5):617-24. doi: 10.2217/fon.12.29. PMID 22646775
- [Background] Blay JY, Serrano C, Heinrich MC, Zalcberg J, Bauer S, Gelderblom H, Schoffski P, Jones RL, Attia S, D'Amato G, Chi P, Reichardt P, Meade J, Shi K, Ruiz-Soto R, George S, von Mehren M. Ripretinib in patients with advanced gastrointestinal stromal tumours (INVICTUS): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Jul;21(7):923-934. doi: 10.1016/S1470-2045(20)30168-6. Epub 2020 Jun 5. PMID 32511981
- [Background] Schuetze SM, Bolejack V, Thomas DG, von Mehren M, Patel S, Samuels B, Choy E, D'Amato G, Staddon AP, Ganjoo KN, Chow WA, Rushing DA, Forscher CA, Priebat DA, Loeb DM, Chugh R, Okuno S, Reinke DK, Baker LH. Association of Dasatinib With Progression-Free Survival Among Patients With Advanced Gastrointestinal Stromal Tumors Resistant to Imatinib. JAMA Oncol. 2018 Jun 1;4(6):814-820. doi: 10.1001/jamaoncol.2018.0601. PMID 29710216
- [Background] Kikuchi H, Hiramatsu Y, Kamiya K, Morita Y, Sakaguchi T, Konno H, Takeuchi H. Surgery for metastatic gastrointestinal stromal tumor: to whom and how to? Transl Gastroenterol Hepatol. 2018 Mar 5;3:14. doi: 10.21037/tgh.2018.02.02. eCollection 2018. PMID 29682621